CLINICAL TRIAL: NCT01975454
Title: A Pilot Study of Teng-Long-Bu-Zhong-Tang Based Herbal Therapy in Combination With Chemotherapy in Patients With Metastatic Colorectal Cancer
Brief Title: Study of TLBZT Based Herbal Therapy Plus Chemotherapy for Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Chongqing Three Gorges Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCM-mCRC; LHYY-11495801300 (Registry Identifier: Longhua Hospital)
Record Dates: First submitted 2013-10-23; First posted 2013-11-04 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2016-10

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic colorectal cancer; Chemotherapy; Traditional Chinese Medicine (TCM); Teng-Long-Bu-Zhong-Tang
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Drug Therapy; Oxaliplatin; Capecitabine; Phytotherapy; Medicine, Chinese Traditional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- chemotherapy (Active Comparator): Patients receive chemotherapy until disease progression or unacceptable toxicity
  Interventions: Drug: Chemotherapy
- Herbal therapy plus chemotherapy (Experimental): Patients receive herbal therapy plus chemotherapy until disease progression or unacceptable toxicity
  Interventions: Drug: Chemotherapy; Drug: Herbal therapy

INTERVENTIONS:
Drug: Chemotherapy — Oxaliplatin (130 mg/m2) was given intravenously (iv) for at least 2 h on day 1; Capecitabine (1000 mg/m2) was given orally, twice daily on days 1-14. Each cycle was 21 days. Cycles were repeated until disease progression or unacceptable toxicity.
  Other Names: Oxaliplatin; Capecitabine
Drug: Herbal therapy — TLBZT based herbal decoction administered orally twice a day
  Other Names: Traditional Chinese Medicine
  Arms: Herbal therapy plus chemotherapy

SUMMARY:
Teng-Long-Bu-Zhong-Tang (TLBZT) is a modern anti-cancer herbal formula. Experimental studies have confirmed the anti-cancer potential of TLBZT against colorectal cancer. This trial will evaluate the safety and efficacy of TLBZT based herbal therapy in combination with chemotherapy in patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
A phase I/II, multicentric,randomized, controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the colon or rectum with non-resectable metastatic disease;
* Ages between 18 and 70 years;
* Measurable lesion;
* Karnofsky Performance Status ≥ 60%;
* Estimated life expectancy of at least 6 months;
* Participants have no major organ dysfunction and chemotherapy contraindications: hemoglobin ≥90g/L, N > 1.5×10^9/L, platelet≥ 100×10^9/L, normal liver and kidney function;
* Informed consent from the patient.

Exclusion Criteria:

* Symptomatic brain metastasis;
* Adjuvant or neo-adjuvant treatment for non-metastatic disease in past 6 months;
* Serious disease of heart, liver, kidney with severe dysfunction;
* Serious complications, such as gastrointestinal tract obstruction and hemorrhage;
* Pregnancy or breast-feeding women;
* Mental or cognitive disorders;
* Be participating other drug trials;
* Who are allergic to the study drug.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-04; Primary Completion 2016-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | 2 months

SECONDARY OUTCOMES:
Overall Survival (OS) | 2 months
Symptoms | 2 months
Adverse events | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Bing Hu, MD, PhD, Study Chair — Shanghai University of Traditional Chinese Medicine; Gang Li, MD, Principal Investigator — Chongqing Three Gorges Central Hospital
Locations (2):
- China (2):
  - Chongqing Three Gorges Central Hospital, Chongqing, Chongqing Municipality
  - Longhua Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Deng S, Hu B, An HM, Du Q, Xu L, Shen KP, Shi XF, Wei MM, Wu Y. Teng-Long-Bu-Zhong-Tang, a Chinese herbal formula, enhances anticancer effects of 5--Fluorouracil in CT26 colon carcinoma. BMC Complement Altern Med. 2013 Jun 8;13:128. doi: 10.1186/1472-6882-13-128. PMID 23758730
- [Background] Hu B, An HM, Shen KP, Du Q. [Senescence-inducing effects of Chinese herbal medicine Tenglong Buzhong Decoction on human colon carcinoma LS-174-T cells and the mechanism]. Zhong Xi Yi Jie He Xue Bao. 2010 Nov;8(11):1048-52. doi: 10.3736/jcim20101108. Chinese. PMID 21078269
- [Background] Hu B, An HM, Shen KP, DU Q. [Effects of Tenglong Buzhong Decoction on proliferation and apoptosis of human colon carcinoma cell line LS174T]. Zhong Xi Yi Jie He Xue Bao. 2010 Jun;8(6):575-80. doi: 10.3736/jcim20100611. Chinese. PMID 20550881